CLINICAL TRIAL: NCT05080920
Title: A Pilot, Randomized, Double Blind, Placebo Controlled Study to Evaluate an Immune System Modulator Nutritional Supplement for the Prevention of Infections in Cancer Patients Receiving Oncologic Treatment During the COVID-19 Pandemia.
Brief Title: Rosmalip® for Cancer Infections Prevention
Acronym: OnCOVInf
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Investigación E Innovación Biomédica Hospital Universitario Infanta Sofia-Henares (Other)
Collaborators: IMDEA Food (Other); Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Enrique Casado Sáenz, Head of Oncology, Fundación Investigación E Innovación Biomédica Hospital Universitario Infanta Sofia-Henares
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Rosmalip®-OnCOVInf
Record Dates: First submitted 2020-10-16; First posted 2021-10-18 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Infections; Covid19; Cancer
MeSH Terms: conditions — Infections; COVID-19; Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants receive Rosmalip® capsule or Placebo tablet matching Rosmalip® orally once daily for 16 weeks.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosmalip® (Experimental): Participants receive Rosmalip® (diterpene phenols 11,25 mg) 1 capsule orally once daily for 16 weeks
  Interventions: Dietary Supplement: Rosmalip®
- Placebo (Placebo Comparator): Participants receive Placebo 1 capsule matching Rosmalip® orally once daily for 16 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Rosmalip® — Nutritional Supplement+Usual Care
  Arms: Rosmalip®
Other: Placebo — Placebo+Usual Care
  Arms: Placebo

SUMMARY:
This study is designed to assess the safety and efficacy of Rosmalip® nutritional supplement compared to placebo in subjects with solid cancer for the prevention of infections including COVID-19.

DETAILED DESCRIPTION:
Cancer patients undergoing oncologic treatments frequently have comorbidities and suffer immunosuppresion, toxicities and exposure to nosocomial pathogens. As a result, they are at increased risk of infections, including COVID-19. It is of utmost importance to find therapies that can prevent infections with as less toxicity as possible. Rosmalip® is a nutritional supplement developed as a molecular nutrition, composed of a rosemary supercritical extract at concentrations approved by EFSA -with in vitro and in vivo antitumor effects that are independent of its antioxidant and anti-inflammatory properties- in a lipidic vehicle that has shown in preclinical and clinical studies to potentiate innate immunity without apparent toxicity. Being a product of easy synthesis its effects on immunity, inflammation and cancer, could be of interest to prevent and ameliorate infections, including COVID-19.

In this pilot study it is hypothesized that Rosmalip® could help to prevent or ameliorate infections, including COVID-19, in oncologic patients under active treatment. Secondarily, it is also hypothesized to have metabolic beneficial effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a solid cancer under active Anticancer Treatment (including Chemotherapy, Immunotherapy, Hormone Therapy, Targeted Therapy)
* Informed consent signature

Exclusion Criteria:

* Allergies to fish
* Vitamin, Antioxidants consumers and who would no accept to stop taking them 1 week before and during the study
* Disphagia
* Bilirrubin higher than 1.5 Upper Normal Limit (UNL)/ Creatinin > 1.5 UNL
* Severe organic dysfunction
* Cardiac dysfunction
* Cholangitis/ Biliary tract obstruction
* Immunodeficiency or Immflamatory disease (HIV, Inflammatory Bowel Disease, Collagenosis)
* Dementia or Psychiatric severe disease
* Pregnancy or Breastfeeding
* Previous diseases that interfere lipid carrier absorption

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of infectious events | 6 months
  Number of infectious events according to International Sepsis Forum Consensus

SECONDARY OUTCOMES:
Number of SARSCoV2 infections | 6 months
  Number of PCR confirmed SARSCoV2 infections
Changes in NLR (neutrophils to lymphocytes ratio). | 6 months
  Evolution of inflammatory markers
Changes in C-reactive protein | 6 months
  Evolution of inflammatory markers
Changes in ferritin | 6 months
  Evolution of inflammatory markers
Changes in transferrin | 6 months
  Evolution of inflammatory markers
Changes in number of peripheral blood mononuclear cells | 6 months
  Evolution of immune profile
Changes in number of CD4 and CD8 lymphocyte populations | 6 months
  Evolution of immune profile
Evolution of Quality of life | 6 months
  Changes is quality of life according to the SF-36 (Short Form Health Survey) questionnaire. The score values goes from 0 to 100 and higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Casado Sáenz, MD, Principal Investigator — Servicio de Oncología. Hospital Infanta Sofía; Ana Ramírez de Molina, PhD, Study Director — IMDEA Food; Guillermo Reglero Rada, PhD, Study Director — CIAL_UAM_CSIC
Locations (1):
- Servicio de Oncología. Hospital Infanta Sofía., San Sebastián de los Reyes, Madrid, Spain

REFERENCES:
- [Background] Mouhid L, Corzo-Martinez M, Torres C, Vazquez L, Reglero G, Fornari T, Ramirez de Molina A. Improving In Vivo Efficacy of Bioactive Molecules: An Overview of Potentially Antitumor Phytochemicals and Currently Available Lipid-Based Delivery Systems. J Oncol. 2017;2017:7351976. doi: 10.1155/2017/7351976. Epub 2017 May 7. PMID 28555156
- [Result] Gomez de Cedron M, Laparra JM, Loria-Kohen V, Molina S, Moreno-Rubio J, Montoya JJ, Torres C, Casado E, Reglero G, Ramirez de Molina A. Tolerability and Safety of a Nutritional Supplement with Potential as Adjuvant in Colorectal Cancer Therapy: A Randomized Trial in Healthy Volunteers. Nutrients. 2019 Aug 24;11(9):2001. doi: 10.3390/nu11092001. PMID 31450563
- [Result] Gonzalez-Vallinas M, Reglero G, Ramirez de Molina A. Rosemary (Rosmarinus officinalis L.) Extract as a Potential Complementary Agent in Anticancer Therapy. Nutr Cancer. 2015;67(8):1221-9. doi: 10.1080/01635581.2015.1082110. Epub 2015 Oct 9. PMID 26452641
- [Result] Gonzalez-Vallinas M, Molina S, Vicente G, Sanchez-Martinez R, Vargas T, Garcia-Risco MR, Fornari T, Reglero G, Ramirez de Molina A. Modulation of estrogen and epidermal growth factor receptors by rosemary extract in breast cancer cells. Electrophoresis. 2014 Jun;35(11):1719-27. doi: 10.1002/elps.201400011. Epub 2014 Mar 20. PMID 24615943
- [Result] Gonzalez-Vallinas M, Molina S, Vicente G, Zarza V, Martin-Hernandez R, Garcia-Risco MR, Fornari T, Reglero G, Ramirez de Molina A. Expression of microRNA-15b and the glycosyltransferase GCNT3 correlates with antitumor efficacy of Rosemary diterpenes in colon and pancreatic cancer. PLoS One. 2014 Jun 3;9(6):e98556. doi: 10.1371/journal.pone.0098556. eCollection 2014. PMID 24892299
- [Result] Gonzalez-Vallinas M, Molina S, Vicente G, de la Cueva A, Vargas T, Santoyo S, Garcia-Risco MR, Fornari T, Reglero G, Ramirez de Molina A. Antitumor effect of 5-fluorouracil is enhanced by rosemary extract in both drug sensitive and resistant colon cancer cells. Pharmacol Res. 2013 Jun;72:61-8. doi: 10.1016/j.phrs.2013.03.010. Epub 2013 Apr 1. PMID 23557932
- [Derived] Gomez de Cedron M, Moreno-Rubio J, de la O Pascual V, Alvarez B, Villarino M, Sereno M, Gomez-Raposo C, Roa S, Lopez Gomez M, Merino-Salvador M, Jimenez-Gordo A, Falagan S, Aguayo C, Zambrana F, Tabares B, Garrido B, Cruz-Gil S, Fernandez Diaz CM, Fernandez LP, Molina S, Crespo MC, Ouahid Y, Montoya JJ, Ramos Ruiz R, Reglero G, Ramirez de Molina A, Casado E. Randomized clinical trial in cancer patients shows immune metabolic effects exerted by formulated bioactive phenolic diterpenes with potential clinical benefits. Front Immunol. 2025 Feb 17;16:1519978. doi: 10.3389/fimmu.2025.1519978. eCollection 2025. PMID 40034703
- [Derived] Bouzas A, Gomez de Cedron M, Colmenarejo G, Laparra-Llopis JM, Moreno-Rubio J, Montoya JJ, Reglero G, Casado E, Tabares B, Sereno M, Ramirez de Molina A. Phenolic diterpenes from Rosemary supercritical extract inhibit non-small cell lung cancer lipid metabolism and synergise with therapeutic drugs in the clinic. Front Oncol. 2022 Nov 9;12:1046369. doi: 10.3389/fonc.2022.1046369. eCollection 2022. PMID 36439419
- See also: ALIBIRD_Therapeutic strategies for precision nutrition in cancer patients — http://www.alibird.org/2020-CM/